CLINICAL TRIAL: NCT07338929
Title: Physical Performance Assessment in Kidney Transplant Evaluation Using the Short Physical Performance Battery (SPPB)
Brief Title: Physical Performance Assessment in Kidney Transplant Evaluation
Acronym: FRAIL-KTx
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, associate professor, University Hospital, Martin
Other Study IDs: TNO FRAIL
Record Dates: First submitted 2025-11-27; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Frailty Syndrome
Keywords: kidney transplantation; chronic kidney diseases; frailty
MeSH Terms: conditions — Frailty; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- kidney transplant recipients: The study will enroll adult patients who are being assessed for kidney transplantation, including those who are deemed suitable and placed on the waiting list (Arm A) and those on dialysis who are considered unsuitable for transplant listing (Arm B).

SUMMARY:
This prospective cohort study investigates physical frailty, assessed by the Short Physical Performance Battery (SPPB), in patients evaluated for kidney transplantation. The study aims to compare SPPB scores before listing, annually during the waiting period, and after transplantation at 6 and 12 months. It also includes a control group of dialysis patients not eligible for transplantation to evaluate differences in physical performance. The goal is to understand how frailty impacts transplant outcomes and patient recovery.

DETAILED DESCRIPTION:
This longitudinal, prospective study focuses on assessing the role of physical frailty in patients undergoing evaluation for kidney transplantation using the Short Physical Performance Battery (SPPB). The study will enroll adult patients who are being assessed for kidney transplantation, including those who are deemed suitable and placed on the waiting list (Arm A) and those on dialysis who are considered unsuitable for transplant listing (Arm B).

Participants will undergo comprehensive SPPB assessments at baseline, during their evaluation process, and subsequently at annual follow-up intervals. For listed patients, the assessments will be performed upon initial evaluation, then annually while on the waiting list, and at 6 and 12 months following transplantation. For patients ineligible for the transplant list and on dialysis, the SPPB will be recorded at baseline and then annually, allowing cross-sectional comparison and understanding of their physical performance trajectory.

The primary objective is to evaluate changes in physical performance over time with the SPPB score, which ranges from 0 to 12. The scores will be used to categorize participants into frail, pre-frail, or non-frail groups, providing insights into the prevalence and evolution of frailty in this population.

Secondary objectives include comparing the baseline and follow-up SPPB scores between the two arms, correlating physical performance with post-transplant outcomes such as graft function and survival, and identifying potential predictors of frailty that could inform prehabilitation interventions.

This study may inform future strategies to optimize physical function in kidney transplant candidates and improve clinical outcomes through targeted interventions addressing physical frailty.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) undergoing evaluation for kidney transplantation.
2. Patients on dialysis.
3. Ability and consent to participate.

Exclusion Criteria:

1. Non-adult patients.
2. Patients unable to provide informed consent.
3. Acute medical conditions prohibiting SPPB assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease undergoing dialysis or pre-transplant evaluation prior to kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
To assess changes in physical performance using SPPB scores before and after kidney transplantation. | 3-5 years
  Characterization of physical performance levels in patients considered for kidney transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Dedinska, prof. MD., PhD., Study Chair — Unievrsity Hospital Martin and Jessenius Faculty of Medicine Comenius University
Locations (1):
- Transplant-nephrology department, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the reported results will be available upon reasonable request from qualified researchers after publication, subject to institutional and ethical approval. Supporting documents (study protocol, statistical analysis plan) may also be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 01/OCT/2025 for 20 years

DOCUMENTS (1):
  • Study Protocol (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT07338929/Prot_000.pdf